CLINICAL TRIAL: NCT00964522
Title: Randomized Trial of the Effectiveness of a Nurse Education and Care Program for Breast Cancer Patients Treated With Chemotherapy
Brief Title: Trial of the Effectiveness of a Nurse Education and Care Program for Breast Cancer Patients Treated With Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Salud Carlos III (Other Government)
Collaborators: Health Service of Andalucia (Other Government)
Responsible Party: Dr. José Manuel Baena Cañada, Hospital Universitario Puerta del Mar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI070141
Record Dates: First submitted 2009-08-17; First posted 2009-08-25 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2010-04

CONDITIONS: Breast Cancer
Keywords: Quality of life; Breast Cancer; Nursing Care; Education; Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): The arm A is the one of standard education and care.
- Nurse education and care program (Active Comparator): The arm B will receive programmed education and care about the chemotherapy by a nurse of the Medical Oncology service before the beginning of the treatment and in each cycle, in a specific nurse consultation.
  Interventions: Other: Nurse education and care program

INTERVENTIONS:
Other: Nurse education and care program — Random allocation of the patients in two arms according to the nursing cares. The arm A is the one of standard education and care. They consist of receiving programmed oral and written information by the specialist before initiating the chemotherapy treatment and before each cycle of treatment. Also, the patients will be able to ask for information to the nurses when they need it. Arm B is the one of experimental education and care. They consist of receiving oral and written information by the specialist before initiating the chemotherapy treatment and before each cycle. In addition, the patients assigned to arm B will receive programmed education and care about the chemotherapy by a Oncology nurse before the beginning of the treatment and in each cycle, in a specific nurse consultation.
  Other Names: Oncology nurse practitioner
  Arms: Nurse education and care program

SUMMARY:
The purpose of this study is to evaluate the effects of a nurse education and care program for patients with breast cancer, in terms of use of the health services, quality of life, satisfaction and security.

Hypothesis:

Nurse education and care program will reduce the use of health resources and will improve the toxicity, quality of life and satisfaction of the patients with breast cancer who initiate chemotherapy.

DETAILED DESCRIPTION:
Design: randomized controlled clinical trial with non-pharmacologic intervention. Subjects and setting of study: patients with breast cancer who initiate adjuvant, neoadjuvant or palliative chemotherapy, in the Day Unit of a University Hospital. Interventions: random allocation of the patients in two arms according to the nursing cares. The arm A is the one of standard education and care. They consist of receiving programmed oral and written information by the specialist in Medical Oncology before initiating the chemotherapy treatment and before each cycle of treatment. Also, the patients will be able to ask for information to the nurses when they need it. Arm B is the one of experimental education and care. They consist of receiving oral and written information by the specialist before initiating the chemotherapy treatment and before each cycle. In addition, the patients assigned to arm B will receive programmed education and care about the chemotherapy by a nurse of the Medical Oncology service before the beginning of the treatment and in each cycle, in a specific nurse consultation. Determinations: use of health resources (not programmed attendance in Primary, Specialist and Emergency care or hospitalisation). Toxicity caused by the chemotherapy. Patients who leave the chemotherapy by serious toxicity. Quality of life measured by means of the EORTC QOL-C30 questionnaire. Satisfaction with the received medical assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer who initiate adjuvant, neoadjuvant or palliative chemotherapy.
* Performance status 0-2 (ECOG).
* Outpatients.
* Normal hematopoietic, hepatic, renal, cardiac and lung functions.
* Must be able to sign the informed consent

Exclusion Criteria:

* Contraindication for chemotherapy
* Inpatients
* Simultaneously radiotherapy and endocrine therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2007-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Use of health resources (not programmed attendance in Primary, Specialist and Emergency care or hospitalisation). | one year

SECONDARY OUTCOMES:
Toxicity. | one year
Quality of life. | one year
Satisfaction | one year

CONTACTS AND LOCATIONS:
Overall Officials: José M. Baena-Cañada, MD; PhD, Study Director — Oncology Unit, Hospital Universitario Puerta del Mar, Cádiz, Spain; Macarena González-Muñoz, Nurse, Principal Investigator — Oncology Unit, Hospital Universitario Puerta del Mar, Cádiz, Spain; Lourdes Solana-Grimaldi, Nurse, Principal Investigator — Oncology Unit, Hospital Universitario Puerta del Mar, Cádiz, Spain; María D. González Piney, Nurse, Principal Investigator — Oncology Unit, Hospital Universitario Puerta del Mar, Cádiz, Spain; Esperanza Arriola-Arellano, MD, Principal Investigator — Oncology Unit, Hospital Universitario Puerta del Mar, Cádiz, Spain
Locations (1):
- Oncology Unit, Hospital Universitario Puerta del Mar, Cadiz, Andalusia, Spain

REFERENCES:
- [Derived] Baena-Canada JM, Estalella-Mendoza S, Gonzalez-Guerrero M, Exposito-Alvarez I, Rosado-Varela P, Benitez-Rodriguez E. [Influence of clinical and biographical factors on the quality of life of women with breast cancer receiving adjuvant chemotherapy]. Rev Calid Asist. 2011 Sep-Oct;26(5):299-305. doi: 10.1016/j.cali.2011.04.005. Epub 2011 Sep 16. Spanish. PMID 21925913